CLINICAL TRIAL: NCT05190458
Title: Evaluation of High Velocity Nasal Insufflation in Management of Respiratory Failure in Patients With Overlap Syndrome.
Acronym: HVNI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Hany Sadek Farag, Resident Doctor at chest department-Assiut University Hospitals, Assiut University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HVNI in Overlap syndrome
Record Dates: First submitted 2021-10-17; First posted 2022-01-13 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Overlap Syndrome; Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Obesity Hypoventilation Syndrome | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive mechanical ventilation (group A) (Other): Patients will be Randomized into 2 subgroups by (1:1) crossover:- Group A will be put on NIMV Group B will be put on HVNI
  Interventions: Other: Non-invasive mechanical ventilation
- High Velocity Nasal Insufflation (group B) (Other): Patients will be Randomized into 2 subgroups by (1:1) crossover:- Group A will be put on NIMV Group B will be put on HVNI
  Interventions: Other: High Velocity Nasal Insufflation

INTERVENTIONS:
Other: High Velocity Nasal Insufflation — High velocity nasal insufflation (HVNI), a form of HFNC that utilizes a small bore nasal cannula to generate higher velocities of gas delivery than HFNC which uses large bore cannula, has the ability to accomplish complete purge of extra thoracic dead space at flow rates of 35 litres/min and may be able to provide ventilatory support in patients with respiratory failure in addition to oxygenation support in patients with overlap syndrome.
  Arms: High Velocity Nasal Insufflation (group B)
Other: Non-invasive mechanical ventilation — Noninvasive ventilation (NIV) refers to the administration of ventilatory support without using an invasive artificial airway (endotracheal tube or tracheostomy tube).
  Arms: Non-invasive mechanical ventilation (group A)

SUMMARY:
High velocity nasal insufflation (HVNI), a form of HFNC that utilizes a small bore nasal cannula to generate higher velocities of gas delivery than HFNC which uses large bore cannula, has the ability to accomplish complete purge of extra thoracic dead space at flow rates of 35 litres/min and may be able to provide ventilatory support in patients with respiratory failure in addition to oxygenation support in patients with overlap syndrome.

This study aims to evaluate the effectiveness of HVNI compared to NIMV in management of respiratory failure in patients with obesity hypoventilation syndrome and overlap syndrome.

DETAILED DESCRIPTION:
Overlap syndrome (OVS) is the concurrence of chronic obstructive pulmonary disease (COPD) and obstructive sleep apnea (OSA), and is associated with poor outcomes.

COPD and obstructive sleep apnoea (OSA) are highly prevalent and different clinical COPD phenotypes that influence the likelihood of comorbid OSA.

The increased lung volumes and low body mass index (BMI) associated with the predominant emphysema phenotype protects against OSA whereas the peripheral oedema and higher BMI often associated with the predominant chronic bronchitis phenotype promote OSA.

The diagnosis of OSA in COPD patients requires clinical awareness and screening questionnaires which may help identify patients for overnight study.

Management of OSA-COPD overlap patients differs from COPD alone and the survival of overlap patients treated with nocturnal positive airway pressure is superior to those untreated.

high flow nasal cannula (HFNC), which delivers heated, humidified oxygen via a nasal cannula at high flow rates of up to 60 L/min, delivering a maximum of 100% oxygen, has been shown to be effective in the treatment of respiratory failure.

High velocity nasal insufflation (HVNI), a form of HFNC that utilizes a small bore nasal cannula to generate higher velocities of gas delivery than HFNC which uses large bore cannula, has the ability to accomplish complete purge of extra thoracic dead space at flow rates of 35 litres/min and may be able to provide ventilatory support in patients with respiratory failure in addition to oxygenation support in patients with obesity hypoventilation syndrome and overlap syndrome.

This study aims to evaluate the effectiveness of HVNI compared to NIMV in management of respiratory failure in patients with overlap syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with respiratory failure in obesity hypoventilation syndrome and overlap syndrome, requiring ICU admission and fulfill criteria of NIMV supplementation (GOLD criteria 2021)
* patients with obesity hypoventilation syndrome and overlap syndrome diagnosed by polysomnogram or through STOP BANG Questionnaire or EPWORTH Sleepness Scale.

Exclusion Criteria:

* Patients less than 18 years old
* Patients with hemodynamic instability
* Patients with central causes of hypercapnic respiratory failure
* Patients with disturbed conscious level
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of HVNI in correction of Acidosis . | Baseline
  Evaluation of the effectiveness of HVNI in correction of Acidosis through measurement of PH via arterial blood gases test (ABG).
Evaluation of HVNI in correction of Hypercapnia. | Baseline
  Evaluation of the effectiveness of HVNI in correction of Hypercapnia through measurement of PCO2 by mmHg via arterial blood gases test (ABG)

SECONDARY OUTCOMES:
Evaluation of HVNI in management of respiratory failure. | Baseline
  Evaluation of the effectiveness of HVNI in management of respiratory failure through measurement of PO2 via arterial blood gases test (ABG)

OTHER OUTCOMES:
Evaluation of HVNI in correction of Hypoxemia. | Baseline
  Evaluation of the effectiveness of HVNI in correction of Hypoxemia through measurement of O2 saturation by percentage % via pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Z El-Abdeen Mohammed, Professor, Principal Investigator — Chest Diseases and Tuberculosis Department-Assiut University Hospitals; Lamiaa H Shaaban, Professor, Study Chair — Chest Diseases and Tuberculosis Department-Assiut University Hospitals; Waleed G Elddin Khaleel, Lecturer, Study Chair — Chest Diseases and Tuberculosis Department-Assiut University Hospitals
Locations (1):
- Respiratory ICU in Assiut University Hospitals, Asyut, Egypt

REFERENCES:
- [Background] Doshi PB, Whittle JS, Dungan G 2nd, Volakis LI, Bublewicz M, Kearney J, Miller TL, Dodge D, Harsch MR, DeBellis R, Chambers KA. The ventilatory effect of high velocity nasal insufflation compared to non-invasive positive-pressure ventilation in the treatment of hypercapneic respiratory failure: A subgroup analysis. Heart Lung. 2020 Sep-Oct;49(5):610-615. doi: 10.1016/j.hrtlng.2020.03.008. Epub 2020 Apr 6. PMID 32273085
- [Background] Doshi P, Whittle JS, Bublewicz M, Kearney J, Ashe T, Graham R, Salazar S, Ellis TW Jr, Maynard D, Dennis R, Tillotson A, Hill M, Granado M, Gordon N, Dunlap C, Spivey S, Miller TL. High-Velocity Nasal Insufflation in the Treatment of Respiratory Failure: A Randomized Clinical Trial. Ann Emerg Med. 2018 Jul;72(1):73-83.e5. doi: 10.1016/j.annemergmed.2017.12.006. Epub 2018 Jan 6. PMID 29310868
- [Background] Poh TY, Mac Aogain M, Chan AK, Yii AC, Yong VF, Tiew PY, Koh MS, Chotirmall SH. Understanding COPD-overlap syndromes. Expert Rev Respir Med. 2017 Apr;11(4):285-298. doi: 10.1080/17476348.2017.1305895. Epub 2017 Mar 24. PMID 28282995
- [Background] Orr JE, Schmickl CN, Edwards BA, DeYoung PN, Brena R, Sun XS, Jain S, Malhotra A, Owens RL. Pathogenesis of obstructive sleep apnea in individuals with the COPD + OSA Overlap syndrome versus OSA alone. Physiol Rep. 2020 Feb;8(3):e14371. doi: 10.14814/phy2.14371. PMID 32061194
- [Background] Masa JF, Pepin JL, Borel JC, Mokhlesi B, Murphy PB, Sanchez-Quiroga MA. Obesity hypoventilation syndrome. Eur Respir Rev. 2019 Mar 14;28(151):180097. doi: 10.1183/16000617.0097-2018. Print 2019 Mar 31. PMID 30872398